CLINICAL TRIAL: NCT01072058
Title: Prospective Evaluation of Heart Function by Echocardiographic Study, Pro-brain Natriuretic Peptide Type B and Troponin T in Patients With Rheumatoid Arthritis and Ankylosing Spondylitis Pre and Post-TNF Blocker
Brief Title: Heart Function in Rheumatoid Arthritis and Ankylosing Spondylitis Pre and Post-TNF Blocker
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Julio Moraes, MD, MD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CapPesq1252/07
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Arthritis, Rheumatoid; Spondylitis, Ankylosing
Keywords: Infliximab; Adalimumab; Etanercept; Heart failure; Diastolic disfunction; TNF blocker; Anti-TNF; Echocardiography; Tissue doppler imaging; Brain Natriuretic Peptide; NT-proBNP
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Heart Failure | interventions — Tumor Necrosis Factor Inhibitors; Infliximab; Adalimumab; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TNF blockers (Other)
  Interventions: Drug: TNF blockers (infliximab, adalimumab, etanercept)

INTERVENTIONS:
Drug: TNF blockers (infliximab, adalimumab, etanercept) — Subjects enrolled, who were eligible to anti-TNF therapy, were evaluated by echocardiography (conventional and tissue doppler imaging)and biomarkers (NT-proBNP and troponin T)at baseline. Then, they were treated with adalimumab 40mg subcutaneously every 2 weeks or infliximab 3 or 5mg/Kg (0, 2 and 6 weeks and thereafter every 8 weeks)or etanercept 50mg subcutaneously every week. And they were re-evaluated with 6, 12, 18 and 24 months from first dose of the TNF blocker .

SUMMARY:
The purpose of this study is to determine possible alterations in cardiac function in patients with Rheumatoid Arthritis and Ankylosing Spondylitis under anti-TNF therapy, without clinical heart disfunction at baseline, using highly sensitive non-invasive methods.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis eligible to receive TNF blockers
* Diagnosis of Ankylosing Spondylitis eligible to receive TNF blockers

Exclusion Criteria:

* Clinical heart failure
* Chagas'disease
* Stable or unstable angina
* Past history of myocardial infarct
* Systemic árterial hypertension (grade 3)
* Valvulopathy
* Chronic kidney disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Development, deterioration ou improvement of subclinical heart dysfunction | 0, 6 ,12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Eloisa S.D.O. Bonfá, MD, PhD, Study Director
Locations (1):
- Rheumatology Division of Hospital das Clínicas da Faculdade de Medicina da Universidade de são PAulo, São Paulo, São Paulo, Brazil